CLINICAL TRIAL: NCT07001839
Title: A Phase Ib Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Preliminary Effectiveness of QLS4131 for Injection in Patients With Systemic Lupus Erythematosus
Brief Title: A Phase Ib Study of QLS4131 in Subjects With Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS4131-201
Record Dates: First submitted 2025-05-25; First posted 2025-06-03 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Systemic Lupus Erythematosus
Keywords: QLS4131; Systemic lupus erythematosus; T cell engager
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS4131 (Experimental): Target dose of each cohort will be administered only once
  Interventions: Drug: QLS4131 for Injection.

INTERVENTIONS:
Drug: QLS4131 for Injection. — Eligible participants will be assigned to 1 of the 9 dose groups ranging from 0.06 μg/kg to 600 μg/kg.

SUMMARY:
The goal of this open label, dose escalation phase 1b clinical trial is to investigate the safety, tolerability, pharmacokinetic, pharmacodynamics, immunogenicity and preliminary clinical efficacy of QLS4131 in subjects with systemic lupus erythematosus (SLE). The main questions it aims to answer are:

* The safety, tolerability and maximum tolerated dose (MTD) of QLS4131 for Injection in participants with SLE.
* The recommended Phase 2 dose (RP2D) of QLS4131 for Injection in participants with SLE.

Participants will be administered different target dose of QLS4131 for Injection only once. A step-up dosing approach will be implemented at high dose level as determined by the safety monitoring committee.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 70 (inclusive);
* Diagnosis of SLE according to the 2019 European League Against Rheumatism/American College of Rheumatology (ACR) Classification Criteria at least 12 weeks or more prior to screening;
* Participants with positive antinuclear antibody (ANA) (≥ 1:80), or positive anti-dsDNA antibody and/or positive anti-Sm antibody at screening;
* Active SLE disease at screening, as demonstrated by a SLEDAI-2K >= 8 at screening, or SLEDAI-2K >= 6 at the presence of low complement and/or positive anti-dsDNA antibodies;
* Current receipt of one or more of the following classes of standard therapies for the treatment of SLE at stable doses: oral corticosteroids, antimalarial agents, and conventional immunosuppressants:

  1. For participants receiving an oral corticosteroid, treatment with ≤40 mg/day prednisone or equivalent, at a dose that has been stable for at least 4 weeks prior to first dose;
  2. For participants receiving an antimalarial, the medication(s) must have been at a stable dose ≥ 4 weeks prior to the first dose;
  3. For participants receiving immunosuppressants, treatment with a single immunosuppressant at a stable dose for ≥ 4 weeks prior to the first dose: conventional immunosuppressants include azathioprine, mycophenolate mofetil, mycophenolic acid, and methotrexate (oral, subcutaneous or intravenous routes).
* Participants who understand and abide by the study procedures, voluntarily participate in this study, and sign the Informed Consent Form in person.

Exclusion Criteria:

* Participants with known intolerance or allergy to the investigational product or drugs that may be used in the study (e.g., Tocilizumab) and any components;
* Participants with active severe active or unstable lupus-associated neuropsychiatric disease;
* Participants with other autoimmune diseases that may affect the efficacy evaluation;
* Participants with poorly controlled hypertension and diabetes;
* Participants with severe lupus nephritis;
* Participants with a history of malignancy within 5 years prior to screening;
* Participants with a previous history of vital organ transplantation;
* Participants who have had opportunistic infections within 12 weeks prior to the first dose;
* Receipt of any CAR-T, CAR-NK or other gene therapy;
* Pregnant or lactating women.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
incidence of treatment emergence adverse events. | Up to 24 weeks]
Recommended Phase 2 Dose | Approximately 24 weeks